CLINICAL TRIAL: NCT05811923
Title: Changes in Metabolic Rate and Perceptual Indicators After Acute Ingestion of Paraxanthine
Acronym: PX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lindenwood University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB-22-30
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Metabolic Syndrome; Caffeine
Keywords: metabolic rate, paraxanthine, caffeine
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Using a randomized, double-blind, placebo-controlled, crossover study design. to ingest one of seven supplement conditions. One condition will be a non-energetic placebo (maltodextrin) while the other six supplemental conditions will be a 200 mg dose of caffeine, 100 mg paraxanthine, 200 mg paraxanthine, 300 mg paraxanthine, a combination of caffeine (200 mg) + paraxanthine (200 mg), and a 200 mg dose of 1-methylxanthine. All supplements will be orally ingested with 8 fluid ounces of cold tap water.
Who Masked: Participant, Investigator
Masking Description: All supplements provided to all research participants containing Caffeine, Paraxanthine, 1-Methylxanthine, or Placebo will be procured and prepared in a similar manner. All supplements are in identical capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator): Maltodextrin placebo capsules
  Interventions: Other: Venous Blood Collection; Other: Resting Metabolic Rate Determination; Other: Mood State; Other: Visual Analog Scales
- 200 mg caffeine (Active Comparator): 200 mg caffeine capsules
  Interventions: Other: Venous Blood Collection; Other: Resting Metabolic Rate Determination; Other: Mood State; Other: Visual Analog Scales
- 100 mg paraxanthine (Experimental): 100 mg paraxanthine capsules
  Interventions: Other: Venous Blood Collection; Other: Resting Metabolic Rate Determination; Other: Mood State; Other: Visual Analog Scales
- 200 mg paraxanthine (Experimental): 200 mg paraxanthine capsules
  Interventions: Other: Venous Blood Collection; Other: Resting Metabolic Rate Determination; Other: Mood State; Other: Visual Analog Scales
- 300 mg paraxanthine (Experimental): 300 mg paraxanthine capsules
  Interventions: Other: Venous Blood Collection; Other: Resting Metabolic Rate Determination; Other: Mood State; Other: Visual Analog Scales
- 200 mg caffeine + 200 mg paraxanthine (Experimental): 200 mg caffeine + 200 mg paraxanthine capsules
  Interventions: Other: Venous Blood Collection; Other: Resting Metabolic Rate Determination; Other: Mood State; Other: Visual Analog Scales
- 200 mg 1-methylxanthine (Experimental): 200 mg 1-methylxanthine capsules
  Interventions: Other: Venous Blood Collection; Other: Resting Metabolic Rate Determination; Other: Mood State; Other: Visual Analog Scales

INTERVENTIONS:
Other: Venous Blood Collection — Within each supplementation condition, study participants will have their venous blood collected on six different occasions: 0, 30, 60, 90, 120, and 180 minutes after ingestion of their assigned study agent. Blood will be collected via a forearm vein using standard phlebotomy techniques using either an indwelling catheter or single venipunctures. All blood samples will be collected into ethylenediaminetetraacetic acid EDTA-coated Vacutainer™ tubes and gently inverted ten times before being centrifuged at 3000 revolutions per minute (rpm) (MegaFuge XFR, Thermo Fisher Scientific, Waltham, MA, USA) at 4oC for 20 minutes. After centrifugation, 400 μl aliquots of plasma will be removed and frozen at -80oC within four hours of collection.
Other: Resting Metabolic Rate Determination — During all study visits and on six occasions during each of the seven experimental conditions (0, 30, 60, 90, 120, and 180 minutes after supplement ingestion), resting metabolic rates will be determined in a thermoneutral laboratory environment.
Other: Mood State — Participants will complete electronic versions of the Profile of Mood States (POMS) questionnaire to evaluate perceptual responses. The Profile of Mood States (POMS) is a 65-item validated scale that uses a 5-point Likert scale with each individual area being scored and summed into profiles for tension, anger, vigor, fatigue, depression, and confusion. Finally, a total mood disturbance score will be calculated by summing all categories and subtracting the vigor score.
Other: Visual Analog Scales — Participants will complete electronic versions of the visual analog (VAS) scale to evaluate perceptual responses. Each VAS scale will be completed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings of focus, anxiety, concentration, energy, restfulness, wakefulness, swagger, confidence, hunger, and appetite. The validity and reliability of VAS to assess fatigue and energy have been previously established (Lee, Hicks, et al. 1991) and our methods have been published elsewhere (Ziegenfuss, Habowski, et al. 2017, Ziegenfuss, Lopez, et al. 2017, Ziegenfuss, Kedia, et al. 2018, Zabriskie, Blumkaitis, et al. 2020).

SUMMARY:
The purpose of this study is to evaluate the acute impact of ingesting individual and combined dosages of caffeine and paraxanthine in comparison to placebo on changes in resting metabolic rate, perceived levels of affect, and markers of lipolysis.

DETAILED DESCRIPTION:
The study will be conducted using a randomized, double-blind, placebo-controlled, crossover study design. Approximately 10 healthy men and 10 healthy women between the ages of 18 - 39 years of age will be recruited to participate in this study. Prior to beginning the study, all participants will sign an IRB-approved informed consent document and complete a healthy history questionnaire to determine study eligibility. All participants will report to the laboratory for all study visits between 0600 - 1000 hours. Prior to each of the seven study visits, participants will be asked to abstain from exercise, tobacco, nicotine, and alcohol for 24 hours and observe an overnight (8 - 10 hours) fast including caffeine. Study visit 1 will be a screening visit where participants will first sign an IRB-approved informed consent document. To determine eligibility, participants will then complete a health and medical history form and have their height and weight assessed along with their resting heart rate and blood pressure. If determined eligible, study participants will allowed to exercise within 24 hours of each study visit. On one occasion prior to study visit 1, study participants will be required to record their food and fluid intake for the three days prior to each study visit and instructed to replicate this diet prior to each visit. To assist in replicating their food intake, participants will be given pre-packaged frozen meals of their choosing. All meals will provide similar amounts of energy, carbohydrates, fats, and proteins. Participants will be instructed to follow an overnight fast whereby no food or fluid with calories will be consumed for the 8 to 10-hour period prior to each study visit. Water intake will be encouraged during this time for appropriate hydration status. Upon arrival for each subsequent study visit, participants will again have their body mass determined and they must be determined to be weight stable (defined as having a body mass within 2% of their previous study visit body mass). Resting heart rate, blood pressure, and body composition will then be assessed (only study visit 2) using a bio-electrical impedance analyzer (BIA). After assessment of body mass, resting heart rate, and resting blood pressure, study participants will donate their first of six venous blood samples. From there, participants will complete a series of assessments evaluating various perceptual indicators using the profile of mood states (POMS) and anchored 100-mm visual analog scales. Finally, participants will then have their resting metabolic rate determined using a metabolic cart. Upon determination of baseline resting metabolic rate, participants will be assigned in a randomized, double-blind, placebo-controlled, crossover fashion to ingest one of seven supplement conditions. One condition will be a non-energetic placebo (maltodextrin) while the other six supplemental conditions will be a 200 mg dose of caffeine, 100 mg paraxanthine, 200 mg paraxanthine, 300 mg paraxanthine, a combination of caffeine (200 mg) + paraxanthine (200 mg), and a 200 mg dose of 1-methylxanthine. All supplements will be orally ingested with 8 fluid ounces of cold tap water. The order of administration for all interventions will be randomized using a random allocation software to ensure randomization and to avoid order effects. After ingestion, participants will complete all assessments in an identical fashion 30, 60, 90, 120, and 180 minutes after ingestion of their assigned supplement. All study visits will take place between 0600 - 1000 hours. It is anticipated that follow-up study visits will be scheduled 3 - 7 days apart from each other after all dietary and exercise controls have been observed.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be between the ages of 18-39 years
* Participants will be healthy and free of disease as determined by evaluation of a - medical history
* All participants will be required to abstain from taking any additional forms of nutritional supplementation (pre-workouts, creatine, beta-alanine, thermogenic supplements, etc.) for four weeks prior to beginning this study and for the entire duration of the study
* Participant's report accumulating at least 30 minutes of moderate exercise 3 days per week
* Currently have a body mass index between 18.5 - 25 kg/m2. Alternatively, individuals with a body mass index between 25 - 30 kg/m2 will be included in the study if body-fat percentage is below 32% for females and 25% for males.
* Not currently restricting calories or completing a dieting program
* As determined through a caffeine intake survey, participants will be moderate caffeine consumers, consuming approximately 200 mg of caffeine per day.

Exclusion Criteria:

* Those individuals less than 18 and greater than 40 years of age will be excluded. Participants younger than 18 are excluded due to necessity of parental consent. Participants greater than 40 years old are excluded due to the known changes that occur with metabolic rate as individuals achieve an age of 40 years or greater
* As indicated on a self-reported medical history, any individual who is currently being treated for or diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic, obesity (defined as body mass index > 30 kg/m2), immune, autoimmune, psychiatric, hematological, neurological, or endocrinological disorder or disease will be excluded.
* Regular (>3 days/week) administration of thermogenic supplements or other weight loss aids in the past 60 days
* Participants not meeting minimum exercise guidelines (30 minutes per day, 3 days per week) or exceeding 8 hours of exercise per week will be excluded
* Daily intake of caffeine doses exceeding 300 mg/day
* Participants who do not or are not willing to abstain from alcohol, nicotine, and caffeine for 12 hours prior to each visit will be excluded
* Participants who do not or are not willing to abstain from exercise for 24 hours prior to each visit will be excluded.
* Participants who do not or are not willing to follow the prescribed dietary control leading up to each exercise bout will be excluded
* Individuals who are pregnant, nursing, or trying to get pregnant

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Rates of resting energy expenditure in response to supplement ingestion | 3 hours
  During all study visits and on six occasions during each of the seven experimental conditions (0, 30, 60, 90, 120, and 180 minutes after supplement ingestion), resting metabolic rates will be determined in a thermoneutral laboratory environment. To complete each assessment, participants will rest supine with a blanket placed over them in an environment free of auditory and visual stimuli. A clear, hard plastic shield with a transparent plastic drape will be placed over the participant's head and shoulder and connected to the metabolic cart to collect all expired gases (oxygen and carbon dioxide). All expired gases will be analyzed using indirect calorimetry (TrueMax 2400 Metabolic Measurement System, ParvoMedics, Sandy, UT, USA) and computed to determine rates of energy expenditure
Total energy expended over a 180-minute time period in response to supplement ingestion | 3 hours
  During all study visits and on six occasions during each of the seven experimental conditions (0, 30, 60, 90, 120, and 180 minutes after supplement ingestion), resting metabolic rates will be determined in a thermoneutral laboratory environment. To complete each assessment, participants will rest supine with a blanket placed over them in an environment free of auditory and visual stimuli. A clear, hard plastic shield with a transparent plastic drape will be placed over the participant's head and shoulder and connected to the metabolic cart to collect all expired gases (oxygen and carbon dioxide). All expired gases will be analyzed using indirect calorimetry (TrueMax 2400 Metabolic Measurement System, ParvoMedics, Sandy, UT, USA) and computed to determine rates of energy expenditure
Perceptual responses of focus, anxiety, concentration, energy, restfulness, wakefulness, swagger and confidence, hunger, and appetite | 3 hours
  Participants will complete electronic versions of the Profile of Mood States (POMS) questionnaire and visual analog (VAS) scale to evaluate perceptual responses. Each VAS scale will be completed using a 100-mm line anchored by "Lowest Possible" and "Highest Possible" to assess subjective ratings of focus, anxiety, concentration, energy, restfulness, wakefulness, swagger, confidence, hunger, and appetite. 0 is lowest level and 5 is highest level.

SECONDARY OUTCOMES:
Rates of carbohydrate and fat oxidation in response to supplement ingestion | 3 hours
  During all study visits and on six occasions during each of the seven experimental conditions (0, 30, 60, 90, 120, and 180 minutes after supplement ingestion), resting metabolic rates will be determined in a thermoneutral laboratory environment. To complete each assessment, participants will rest supine with a blanket placed over them in an environment free of auditory and visual stimuli. A clear, hard plastic shield with a transparent plastic drape will be placed over the participant's head and shoulder and connected to the metabolic cart to collect all expired gases (oxygen and carbon dioxide). All expired gases will be analyzed using indirect calorimetry (TrueMax 2400 Metabolic Measurement System, ParvoMedics, Sandy, UT, USA) and computed to determine rates of carbohydrate and fat oxidation in response to supplement ingestion
Plasma concentrations of glycerol and free fatty acids after supplement ingestion | 3 hours
  The collected blood will be analyzed using a hand-held glucose analyzer and fasting will be considered confirmed if glucose is < 110 mg/dL. Within each supplementation condition, study participants will have their venous blood collected on six different occasions: 0, 30, 60, 90, 120, and 180 minutes after ingestion of their assigned study agent

OTHER OUTCOMES:
Changes in resting heart rate in response to supplement ingestion. | 3 hours
  Resting heart rate (bpm) measured at all 6 time points over 180 minutes
Changes in systolic blood pressure (mmHg) in response to supplement ingestion. | 3 hours
  Systolic blood pressure (mmHg) are measured at all 6 time points across 180 minutes
Changes in diastolic blood pressure (mmHg) in response to supplement ingestion. | 3 hours
  Diastolic blood pressure (mmHg) are measured at all 6 time points across 180 minutes
Changes in adverse events | 3 hours
  Adverse events are self-reported at all study visits and all time-points

CONTACTS AND LOCATIONS:
Overall Officials: Chad M Kerksick, PhD, Principal Investigator — Lindenwood University
Locations (1):
- Exercise and Performance Nutrition Laboratory, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: No